CLINICAL TRIAL: NCT01105260
Title: Effects of an Early Wheelchair Reconditionong Program on Functional Independence in Spinal Cord-inured Individuals
Status: Terminated | Type: Observational
Why Stopped: Difficulty to include patients
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 0901040; 2009-A00866-51 (Other: AFSSAPS)
Record Dates: First submitted 2010-03-23; First posted 2010-04-16 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Spinal Cord Injuries
Keywords: early reconditioning program; spinal cord injury; early rehabilitation; wheelchair
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- control: group with classical rehabilitation program
- training: group with an 8 weeks interval training program on wheelchair independence

SUMMARY:
Reconditioning program during the chronic phase of the spinal cord-injury is well known for its beneficial effects, but there is no investigation in early rehabilitation consequences. Nevertheless, it may be justified : to increase oxygen uptake; to decrease the risks of medical complications; or to improve the mobility. The restrictive autonomy is due to different factors: firstly wheelchair users reduce their movement because they need technical or human help to achieve transfers; and secondly, locomotion is performed by the upper limbs. Without specific practice, the upper limbs mechanical and physiological properties do not permit exercises that are long and intense. Then, the purpose of this research is to evaluate the effects of an 8 weeks interval training program on wheelchair independance during inpatient early rehabilitation for spinal cord injury (3 to 6 months post injury) compared to a control group (classical rehabilitation program in a physical medicine and rehabilitation department).

ELIGIBILITY:
Inclusion Criteria:

* Acute spinal cord injury (SCI) from trauma , medical or surgical pathology at levels between C7 and L1.
* Categories A or B as defined by the American Spinal Injury Association (ASIA) Impairment Scale
* Male or female
* 18 to 60 years old.
* No ability to walk independently with or without an assistive device
* 3 to 6 months post-SCI in early phase of rehabilitation in a physical medicine and rehabilitation unit.
* Subject affiliated to a social security regime and registered at the healthcare department
* Written informed consent obtained from each subject

Exclusion Criteria:

* Symptomatic syringomyelia that may complicate the evaluation procedures
* Disabled pathology before the SCI
* Cardiopulmonary disease, degenerative disorders, upper limb disorders, bones inury or other significant medical complications that would prohibit or alter compliance with a wheelchair training protocol.
* Psychological incapacity to follow a training protocol during 8 weeks.
* Surgery or intrathecal injection planned.
* Reject to give written informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with acute spinal cord injury (SCI) from trauma, medical or surgical pathology at levels between C7 and L1
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
wheelchair independence and mobility | inclusion and 6 month
  adapted 6-minutes walk test (maximal distance ran in 6 minutes with patient's personal wheelchair) crossing a 5% slope functional independence measure (FIM) quality of life

SECONDARY OUTCOMES:
Cardiovascular parameters | inclusion and 6 month
  Maximal exercise test (maximal oxygen uptake, maximal tolerated power (MTP), ventilatory threshold (VS), maximal heart rate, blood pressure, blood lactate) Three exercise tests to exhaustion (work rate fixed at 90, 100 and 110 % MTP, to determine the critical power (power which can be sustained without fatigue)
Biomechanic parameters during manuel wheelchair propulsion | inclusion and 6 month
  Push phases push frequency total cycle time

CONTACTS AND LOCATIONS:
Overall Officials: Paul Calmels, MD, Principal Investigator — CHU de Saint-Etienne
Locations (8):
- France (8):
  - CHU Besançon, Besançon
  - Centre de Rééducation de la Tour de Gassie, Bruges
  - Groupe Hospitalier Raymond Poincaré - APHP, Garches
  - Service MPR des Kermes - Hôpital René Sabran, Giens
  - Centre mutualiste neurologique Propara, Montpellier
  - CHU Nantes, Nantes
  - Centre mutualiste de Rééducation et de Réadaptation Fonctionnelles de Kerpape, Ploemeur
  - Centre de Réadaptation fonctionnelle - UGECAM, Strasbourg